CLINICAL TRIAL: NCT04093050
Title: A Phase 1, Open-Label, Two-Arm, Parallel-Group, Pharmacokinetic Study on Plasma Clearance of Vasopressin in Healthy Volunteers
Brief Title: Safety and Pharmacokinetics of Vasopressin in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Endo Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PS4229-101
Record Dates: First submitted 2019-09-16; First posted 2019-09-17 (Actual); Last update posted 2021-05-19 (Actual); Status verified 2021-04

CONDITIONS: Healthy Volunteer Safety Study

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- TT Genotype (Experimental)
  Interventions: Drug: Vasostrict Injectable Product
- AA/AT Genotype (Experimental)
  Interventions: Drug: Vasostrict Injectable Product

INTERVENTIONS:
Drug: Vasostrict Injectable Product — Vasostrict® (vasopressin injection, USP)

SUMMARY:
Open-label Phase I pharmacokinetic (PK) study of Vasostrict® (vasopressin injection, USP) in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

1. Signed the informed consent form (ICF) approved by an institutional review board (IRB).
2. Determined to have genotype TT, AA, or AT.
3. Weighs at least 50 kg and not more than 100 kg.
4. If female, must be surgically sterile for at least 6 months prior to screening, post-menopausal for at least 1 year, using adequate contraception, have a vasectomized partner or abstinent.
5. Participant is in good physical health as determined by the investigator, based on physical examination, medical history, 12-lead ECG, vital signs, and clinical laboratory tests.
6. Participant is willing and able to comply with all aspects of the protocol, including the diet and medication restrictions.

Exclusion Criteria:

1. If female, breastfeeding or pregnant.
2. Use of any prescription or over-the-counter drugs.
3. Clinical laboratory test results outside laboratory normal range that are determined by the investigator to be clinically significant.
4. Creatinine clearance <90 mL/min (estimated by Cockcroft-Gault formula).
5. Pulse rate ≤50 or ≥100 bpm, systolic blood pressure ≤90 or ≥140 mmHg, diastolic blood pressure ≤60 or ≥90 mmHg or a history of hypertension, recurrent hypotensive events, or known orthostatic hypotension.
6. ECG abnormalities (PR >200 msec; QRS complex >120 msec; QT interval corrected for heart rate using Fridericia's formula [QTcF] interval >450 msec if male and >470 msec if female, or history of clinically significant ECG abnormalities (such as cardiac arrhythmia, familial long QT syndrome, or previous torsade de pointes).
7. History of diabetes insipidus, syndrome of inappropriate antidiuretic hormone secretion, or any other disorder associated with fluid or sodium imbalance.
8. History or evidence of any clinically significant surgical or medical condition (eg, cardiovascular, gastrointestinal, endocrine, hematologic, hepatic, immunologic, metabolic, urologic, pulmonary, neurologic, psychiatric, dermatologic, renal, and/or another major disease or malignancy) that would be anticipated, in the opinion of the investigator, to compromise participant safety or PK evaluation.
9. Known allergy or hypersensitivity to 8-L-arginine vasopressin or chlorobutanol.
10. Clinically significant history of allergic conditions (including drug allergies, asthma, eczema, or anaphylactic reactions, but excluding untreated, asymptomatic seasonal allergies), as judged by the investigator.
11. History of or current infection with hepatitis B virus, hepatitis C virus, or human immunodeficiency virus.
12. Use of tobacco- or nicotine-containing products in the 6 months prior or intent to smoke during the study. Smoking status will be confirmed by negative urine cotinine test.
13. Consumption of more than 21 units (males) or more than 14 units (females) of alcohol per week (1 unit = 10 g pure alcohol or 250 mL of beer [5%], 35 mL of spirits [35%], or 100 mL of wine [12%]). Alcohol use is prohibited from 72 hours prior to admission on Day -2 until discharge from clinical unit.
14. History of chronic drug or alcohol abuse in the last 4 years. Lack of abuse will be confirmed by urine screens for alcohol and drugs of abuse (amphetamines, barbiturates, benzodiazepines, cannabinoids, cocaine metabolites, methamphetamines, methylenedioxymethamphetamine, and opiates [including heroin, codeine, and oxycodone]).
15. Participation in a clinical trial of an investigational drug within the 30 days prior to admission on Day -2.
16. Significant blood loss or donation (≥500 mL within the 30 days prior to admission on Day -2).
17. Is an employee or the close relative of an employee of the sponsor or clinical unit.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2019-10-10 (Actual); Primary Completion 2021-04-08 (Actual); Study Completion 2021-04-11 (Actual)

PRIMARY OUTCOMES:
Plasma Clearance of vasopressin following IV administration in participants with TT genotype versus AA/AT genotype | 15 days

CONTACTS AND LOCATIONS:
Overall Officials: Shannon Dalton, Study Director — Endo Pharmaceuticals
Locations (2):
- United States (2):
  - Endo Clinical Trial Site #2, Orlando, Florida
  - Endo Clinical Trial Site #1, Austin, Texas

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP